CLINICAL TRIAL: NCT00394355
Title: Comparative Study of the Effect of Two Doses of Mometasone Furoate Dry Powder Inhaler 200 mcg and 400 mcg QD PM, Fluticasone Propionate 250 mcg BID, and Montelukast 10 mg QD PM, on Bone Mineral Density in Adults With Asthma
Brief Title: Effects of Mometasone Furoate Dry Powder Inhaler, Fluticasone Propionate, and Montelukast on Bone Mineral Density in Asthmatics (Study P03418)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P03418; Doc ID: 3387777;; EUDRACT No: 2004-002930-21;
Record Dates: First submitted 2006-10-31; First posted 2006-11-01 (Estimated); Results first posted 2011-03-07 (Estimated); Last update posted 2024-05-22 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate; Fluticasone; montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Experimental): MF DPI 400 mcg once a day (QD) in the evening (PM)
  Interventions: Drug: mometasone furoate dry powder inhaler
- Group 2 (Experimental): MF DPI 200 mcg QD PM
  Interventions: Drug: mometasone furoate dry powder inhaler
- Group 3 (Active Comparator): Fluticasone propionate (FP) metered dose inhaler (MDI) 250 mcg twice a day (BID)
  Interventions: Drug: fluticasone propionate hydrofluoroalkane (HFA)
- Group 4 (Active Comparator): ML 10 mg QD PM
  Interventions: Drug: montelukast

INTERVENTIONS:
Drug: mometasone furoate dry powder inhaler — 400 mcg MF DPI via a breath-actuated, dry-powder inhaler and a placebo tablet given by mouth once daily in the evening for 1 year.
  Other Names: Asmanex
  Arms: Group 1
Drug: mometasone furoate dry powder inhaler — 200 mcg MF DPI via a breath-actuated, dry-powder inhaler and a placebo tablet given by mouth once daily in the evening for 1 year.
  Other Names: Asmanex
  Arms: Group 2
Drug: fluticasone propionate hydrofluoroalkane (HFA) — 250 mcg FP HFA given twice a day via a metered-dose inhaler and a placebo tablet given once daily in the evening for 1 year
  Other Names: Flovent HFA
  Arms: Group 3
Drug: montelukast — 10 mg given once daily in the evening by mouth for 1 year.
  Other Names: Singulair
  Arms: Group 4

SUMMARY:
This is a randomized, multi-center, parallel-group, active-controlled, double-blind study evaluating the effects of mometasone furoate (MF) dry powder inhaler (DPI) on bone mineral density (BMD) in subjects with asthma. The mean percent change in lumbar spine BMD from the averaged baseline value (the average of the two scan results prior to treatment) to the endpoint of treatment time point (the average of the last two valid post-baseline scan results during treatment) for the comparison of MF DPI 400 mcg daily in the evening versus montelukast (ML) 10 mg daily in the evening.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent, adhere to schedules.
* Inform usual treating medical doctor (MD) of study participation.
* Female 18 to 40, male 18 to 50, any race.
* >=3-month asthma history.
* Never treated with inhaled corticosteroids (ICS) for asthma or not have taken ICS for ≥3 months prior to Screening.
* Prebronchodilator forced expiratory volume (liters) in 1 second (FEV1) >=60% & <=90% predicted at both Screening & Baseline, when all restricted medications withheld.
* Prior to randomization, demonstrate increase in absolute FEV1 of >=12%, with absolute volume increase of >=200 mL, after reversibility testing.
* Lab tests normal/acceptable to investigator/sponsor. Electrocardiogram (ECG) performed at screening or <30 days of screening normal/acceptable to investigator. Chest x-ray performed at screening or <12 months of screening normal/acceptable to investigator.
* 25-hydroxy vitamin D level >=15 ng/mL. If <15, re-tested after taking calcium plus vitamin D for 4 weeks.
* Free of significant disease (other than asthma) known to affect bone mineral metabolism including renal disease, unstable hyperthyroidism or other endocrinopathies, Paget's disease, osteoporosis, malabsorption, or others that could interfere with study evaluations (eg scoliosis, metal pins, calcification in spine/femur).
* Women of childbearing potential must use birth control. Includes: hormonal contraceptive, intra-uterine device (IUD); condom in combination with spermicide; monogamous relationship with male who had vasectomy or is using condom. Started method ≥3 months prior to Screening (exception condom), & agree to continue for duration. Women who are not currently sexually active must agree/consent to using double-barrier method if become active. Females must have negative serum pregnancy test at Screening.
* 2 valid scans, as confirmed by local dual energy x-ray absorptiometry (DXA) center, for lumbar spine, left total femur, & femoral neck prior to randomization. Valid scans will be 2 scans of same region, performed on same day, that agree within 5% & scans are technically satisfactory (eg correct scan mode, no artifacts present, correct region).

Exclusion Criteria:

* >12 inhalations/day of salbutamol on 2 consecutive days between Screening & Baseline.
* Increase/decrease in FEV1 of >=20% between Screening & Baseline.
* Treated with methotrexate, cyclosporin, gold, or other cytotoxic agents, for asthma or concurrent condition within last 3 months.
* Pipe/cigar smoking history.
* Smoker/ex-smoker who smoked within previous year or has smoking history ≥10 pack-years.
* Upper/lower respiratory tract infection within 2 weeks prior to Screening & Baseline. Can be rescheduled.
* >14 days of oral steroids within previous 12 months or required burst of systemic steroids within previous month.
* Ever required ventilator support for respiratory failure secondary to asthma.
* Treated in emergency room (ER) for asthma exacerbation or admitted to hospital for management of airway obstruction on 1 occasion in last 3 months or on >=2 occasions within last 6 months.
* Chronic bronchitis, bronchiectasis, emphysema or cystic fibrosis.
* Participated in study within last 30 days.
* Allergic to/intolerant of ICS, beta-agonists, or drugs/excipients in study.
* Average of 2 lumbar spine (L1-L4) scans at Screening is >2 standard deviations below normal.
* Condition that might affect ability to ambulate normally, (ie major surgical procedure). Condition that may interfere with BMD measurement.
* History of renal, hepatic, cardiovascular, metabolic, neurologic, hematologic, respiratory, gastrointestinal, cerebrovascular, or other which could interfere with study or require treatment which might interfere (eg calcium urolithiasis or absorptive hypercalcuria, insulin dependent diabetes, cancer within last 10 years (except basal cell carcinoma), active hepatitis, coronary artery disease, stroke, rheumatoid arthritis, human immunodeficiency virus (HIV), or respiratory conditions such as chronic obstructive pulmonary disease (COPD), chronic bronchitis, cystic fibrosis. Others which are well-controlled & stable (eg hypertension, arrhythmia, subjects on stable thyroid hormone replacement for at least 3 months whose thyroid stimulating hormone (TSH) levels are normal) may be allowed.
* Treated within last year with drug known to interfere with bone metabolism including: bisphosphonates, estrogens such as depot injectables (estrogens used in oral combined hormonal contraceptives are allowed if dose is stable throughout), high-dose fluoride, & thyroid replacement hormones (if not stabilized).
* History &/or presence of intraocular pressure in either eye >=22 mm Hg, glaucoma, &/or posterior subcapsular cataracts. History &/or presence of nuclear cataract or undergone bilateral lens extraction may be eligible.
* The subject has undergone incisional or intraocular surgery in which the natural lens is still present in the eye.
* The subject has a history of penetrating trauma to both eyes.
* The subject has one or more of the following lens opacities classification system version III (LOCS III) grades at screening: nuclear opalescence (NO) >=3.0, nuclear color (NC) >=3.0, cortical (C) >=2.0, posterior (P) >=0.5.
* Pregnant, breast-feeding, or postmenopausal women. Amenorrhea >6 months will be excluded (exception hysterectomy). Bilateral oophorectomy excluded.
* Relevant abnormal Baseline vital sign.
* Body mass index (BMI) >35 kg/m2.
* HIV positive (testing not performed).
* Alcoholic or illicit drug abuser.
* Evidence of oropharyngeal candidiasis at Baseline with or without treatment. If evidence at Screening, may be treated as appropriate & visit can be scheduled upon resolution. If evidence at Baseline Visit, may be treated as appropriate & visit can be rescheduled upon resolution.
* Normal sleep/wake cycle is inverted (eg night shift workers).
* Taken restricted medications prior to Screening.
* Cannot adhere to prohibited & permitted concomitant medications.
* No subject may participate in this same study at another site or simultaneously in any other study.
* No person directly associated with administration of study may participate.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 566 (Actual)
Dates: Start 2006-09; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Maspero J, Backer V, Yao R, Staudinger H, Teper A. Effects of mometasone, fluticasone, and montelukast on bone mineral density in adults with asthma. J Allergy Clin Immunol Pract. 2013 Nov-Dec;1(6):649-55.e1. doi: 10.1016/j.jaip.2013.07.011. Epub 2013 Oct 8. PMID 24565713

RESULTS

PARTICIPANT FLOW:
Groups:
- MF DPI 200 mcg QD PM: Mometasone furoate (MF) dry powder inhaler (DPI) 200 mcg once daily (QD) in the evening (PM) for 1 year
- MF DPI 400 mcg QD PM: MF DPI 400 mcg QD PM for 1 year
- FP MDI 250 mcg BID: Fluticasone proprionate (FP) metered dose inhaler (MDI) 250 mcg twice daily (BID) for 1 year
- ML 10 mg QD PM: Montelukast (ML) 10 mg QD PM for 1 year
Period: Overall Study
Arm/Group | MF DPI 200 mcg QD PM | MF DPI 400 mcg QD PM | FP MDI 250 mcg BID | ML 10 mg QD PM
Started | 140 | 137 | 147 | 142
Completed | 105 | 103 | 109 | 111
Not Completed | 35 | 34 | 38 | 31
Not completed — Adverse Event | 10 | 6 | 7 | 8
Not completed — Did not meet protocol eligibility | 1 | 5 | 4 | 2
Not completed — Subject withdrawal - unrelated to drug | 12 | 14 | 10 | 6
Not completed — Subject withdrawal - related to drug | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 7 | 5 | 4 | 3
Not completed — Noncompliance with protocol | 4 | 3 | 10 | 8
Not completed — Administrative | 0 | 1 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MF DPI 200 mcg QD PM | MF DPI 400 mcg QD PM | FP MDI 250 mcg BID | ML 10 mg QD PM | Total
Number analyzed (Participants) | 140 | 137 | 147 | 142 | 566
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.7 (7.8) | 29.8 (8.1) | 28.2 (6.9) | 28.2 (7.1) | 29.0 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 90 | 90 | 88 | 359
  Male | 49 | 47 | 57 | 54 | 207

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in Lumbar Spine Bone Mineral Density (BMD) From the Averaged Baseline Value to the Endpoint of Treatment Time Point
Description: The averaged baseline value is the average of the two scan results prior to treatment. The endpoint of treatment time point is the average of the last two valid post baseline BMD scans during the treatment period carried forward.
Time Frame: Baseline and up to ~ one year of treatment
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: percentage of BMD
Arm/Group | MF DPI 200 mcg QD PM | MF DPI 400 mcg QD PM | FP MDI 250 mcg BID | ML 10 mg QD PM
Number analyzed (Participants) | 117 | 121 | 131 | 127
percentage of BMD | 0.7 (2.56) | 0.9 (2.56) | 1.1 (2.56) | 1.2 (2.56)
Statistical Analysis 1: Comparison: MF DPI 400 mcg QD PM vs ML 10 mg QD PM; Least squares mean percent changes were obtained from the two-way analysis of variance (ANOVA) model with treatment and BMD scan center effects. Results shown use percent change as a response. Pooled Standard deviation from the ANOVA model with treatment effects; Test type: Superiority or Other; p = 0.261, ANOVA
Statistical Analysis 2: Comparison: FP MDI 250 mcg BID vs ML 10 mg QD PM; Least squares mean percent changes were obtained from the two-way ANOVA model with treatment and BMD scan center effects. Results shown use percent change as a response. Pooled Standard deviation from the ANOVA model with treatment effects; Test type: Superiority or Other; p = 0.644, ANOVA

2. Secondary Outcome: Mean Percent Change in the Left Total Femur From the Averaged Baseline Value to the Averaged Value at the Endpoint of Treatment Time Point
Description: as for outcome 1
Time Frame: Baseline and up to ~ one year of treatment
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: percentage of BMD
Arm/Group | MF DPI 200 mcg QD PM | MF DPI 400 mcg QD PM | FP MDI 250 mcg BID | ML 10 mg QD PM
Number analyzed (Participants) | 117 | 121 | 130 | 127
percentage of BMD | 0.3 (2.00) | 0.2 (2.00) | 0.2 (2.00) | 0.5 (2.00)
Statistical Analysis 1: Comparison: MF DPI 400 mcg QD PM vs ML 10 mg QD PM; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.359, ANOVA
Statistical Analysis 2: Comparison: FP MDI 250 mcg BID vs ML 10 mg QD PM; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.390, ANOVA

3. Secondary Outcome: Mean Percent Change in the Femoral Neck BMD From the Averaged Baseline Value to the Averaged Value at the Endpoint of Treatment Time Point
Description: as for outcome 1
Time Frame: Baseline and up to ~ one year of treatment
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: percentage of BMD
Arm/Group | MF DPI 200 mcg QD PM | MF DPI 400 mcg QD PM | FP MDI 250 mcg BID | ML 10 mg QD PM
Number analyzed (Participants) | 117 | 121 | 130 | 127
percentage of BMD | -0.2 (3.17) | 0.4 (3.17) | -0.4 (3.17) | -0.2 (3.17)
Statistical Analysis 1: Comparison: MF DPI 400 mcg QD PM vs ML 10 mg QD PM; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.169, ANOVA
Statistical Analysis 2: Comparison: FP MDI 250 mcg BID vs ML 10 mg QD PM; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.526, ANOVA

4. Secondary Outcome: Summary of Change From Baseline to Endpoint in FEV1 (Forced Expiratory Volume in One Second).
Description: Mean percent change from Baseline (the last non-missing value prior to treatment) in pulmonary function test FEV1 from in-office visits and at Endpoint (last non-missing postbaseline value carried forward)
Time Frame: Baseline and up to ~ one year of treatment
Measure: Mean (Standard Deviation); unit: percentage of FEV1
Arm/Group | MF DPI 200 mcg QD PM | MF DPI 400 mcg QD PM | FP MDI 250 mcg BID | ML 10 mg QD PM
Number analyzed (Participants) | 140 | 136 | 146 | 141
percentage of FEV1 | 0.29 (0.43) | 0.38 (0.43) | 0.31 (0.43) | 0.19 (0.43)
Statistical Analysis 1: Comparison: MF DPI 400 mcg QD PM vs ML 10 mg QD PM; Least square means and Pstd (pooled standard deviations) are obtained from the ANOVA model with treatment effects; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: FP MDI 250 mcg BID vs ML 10 mg QD PM; Least square means and Pstd (pooled standard deviations) are obtained from the ANOVA model with treatment effects; Test type: Superiority or Other; p = 0.023, ANOVA

ADVERSE EVENTS:
Arm/Group | MF DPI 200 mcg QD PM | MF DPI 400 mcg QD PM | FP MDI 250 mcg BID | ML 10 mg QD PM
Serious Adverse Events (participants affected / at risk) | 5/140 | 2/137 | 4/147 | 8/142
Other Adverse Events (participants affected / at risk) | 61/140 | 69/137 | 75/147 | 64/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MF DPI 200 mcg QD PM (N=140) | MF DPI 400 mcg QD PM (N=137) | FP MDI 250 mcg BID (N=147) | ML 10 mg QD PM (N=142)
Lenticular opacities (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Keratitis herpetic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Victim of homicide (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MF DPI 200 mcg QD PM (N=140) | MF DPI 400 mcg QD PM (N=137) | FP MDI 250 mcg BID (N=147) | ML 10 mg QD PM (N=142)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 4 (5) | 8 (28) | 6 (7)
Dyspepsia (Gastrointestinal disorders) | 4 (12) | 7 (8) | 2 (3) | 2 (3)
Bronchitis (Infections and infestations) | 3 (4) | 10 (12) | 7 (8) | 10 (13)
Influenza (Infections and infestations) | 14 (16) | 10 (15) | 11 (13) | 13 (19)
Nasopharyngitis (Infections and infestations) | 16 (29) | 27 (45) | 26 (40) | 23 (32)
Pharyngitis (Infections and infestations) | 17 (19) | 14 (19) | 11 (15) | 12 (15)
Rhinitis (Infections and infestations) | 3 (4) | 6 (28) | 3 (6) | 9 (21)
Upper respiratory tract infection (Infections and infestations) | 6 (9) | 10 (15) | 7 (7) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 10 (14) | 9 (11) | 4 (6)
Headache (Nervous system disorders) | 22 (55) | 18 (38) | 19 (37) | 21 (93)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 7 (12) | 9 (14) | 11 (35) | 7 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigator (PI) agrees not to publish or publicly present any interim results of the study without prior written consent of the sponsor. The PI further agrees to provide to the sponsor, 30 days prior to submission, review copies for publication that report any study results. The sponsor has the right to review and comment. If the parties disagree, PI agrees to meet with the sponsor, prior to submission for publication, to discuss and resolve any such issues or disagreement.